CLINICAL TRIAL: NCT00249977
Title: Phase I Study Of Capecitabine in Combination With Cisplatin and Irinotecan in Patients With Advanced Malignancies.
Brief Title: Phase I Study of Capecitabine in Combination With Cisplatin and Irinotecan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Claire Verschraegen, M.D.; Principal Investigator, University of New Mexio - CRTC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103C
Record Dates: First submitted 2005-11-02; First posted 2005-11-07 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-10

CONDITIONS: Solid Tumors; Cancer
Keywords: Phase I; solid tumors; DNA repair
MeSH Terms: conditions — Neoplasms | interventions — Capecitabine; Cisplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Capecitabine in Combination with Cisplatin and Irinotecan — Cisplatin 50 mg/m2 on day 1 (course 1) or day 11 (subsequent courses) Irinotecan 50 mg/m2 on day 1, 8, and 15 (course 1) or day 11, 18 and 25 (subsequent courses).
  Capecitabine will be administered from day 1 to day 10 PO starting on course 2.

SUMMARY:
1. To determine the safety and feasibility of administering Capecitabine with the combination of Cisplatin and Irinotecan.
2. To determine the Phase II recommended dose and toxicity profile of Capecitabine with the combination of Cisplatin and Irinotecan.
3. To study the biologic effect of pyrimidine inhibition on DNA repair after camptothecin therapy.

DETAILED DESCRIPTION:
RATIONALE: Many studies have tested the combination of cisplatin and irinotecan. Side effects have been well described. The two drugs are synergistic.

The standard of care for colon cancer is the combination of 5-FU, leucovorin and irinotecan (Saltz regimen). Recently, oxaliplatin has been introduced for the treatment of colon cancer. Combination of oxaliplatin with 5FU (Folfox4) have shown comparable activity to the Saltz regimen. Furthermore, one author recently published on the triple combination of oxaliplatin, 5FU and irinotecan, with impressive clinical activity in colon cancer.

There is some evidence that 5FU impairs DNA repair. One of the putative resistance mechanism to topoisomerase I inhibitors is increased DNA repair. We therefore hypothesize that inhibition of DNA repair by capecitabine may increase the activity of the combination of cisplatin and irinotecan.

This study is open to all patients with solid tumor who have failed a line of chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* All patients, 18 years of age or older, with incurable advanced cancer for whom there is no effective therapy are eligible.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of > 1,500 or cells/mm3 and platelet count >100,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 1.5 x upper limit of normal.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.
* Patients whose cancer progressed while receiving 5-FU, cisplatin or irinotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-04; Primary Completion 2007-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety/feasibility of Capecitabine with the combination of Cisplatin and Irinotecan. To determine the Phase II recommended dose and toxicity profile of Capecitabine with the combination of Cisplatin and Irinotecan. | Progressing disease or unacceptable toxicities

SECONDARY OUTCOMES:
To study the biologic effect of pyrimidine inhibition on DNA repair after camptothecin therapy. | disease progression, unacceptable toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Claire F Verschraegen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States